CLINICAL TRIAL: NCT02057640
Title: A Phase I/II Study of MLN9708 (Ixazomib) in Combination With Panobinostat and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: MLN9708 (Ixazomib) in Combination With Panobinostat and Dexamethasone in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jason Valent (Other)
Responsible Party: Sponsor-Investigator, Jason Valent, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4A13
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma; Kahler Disease; Plasma-Cell Myeloma; Myelomatosis
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat; Dexamethasone; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination therapy: Panobinostat, dexamethasone, MLN9708 (Experimental): Panobinostat: 20mg, on day 1, 3, 5, 15, 17, 19, 28 Dexamethasone: 20mg, on day 1, 2, 8, 9, 15, 16, 28 MLN9708: 4mg on day 1, 8, 15, 28
  Interventions: Drug: Panobinostat; Drug: Dexamethasone; Drug: MLN9708

INTERVENTIONS:
Drug: Panobinostat — 20mg, on day 1, 3, 5, 15, 17, 19, 28
Drug: Dexamethasone — 20mg, on day 1, 2, 8, 9, 15, 16, 28
Drug: MLN9708 — 4mg on day 1, 8, 15, 28
  Other Names: Ixazomib

SUMMARY:
This study will look at the safety and tolerability of the new drug MLN9708 in combination with the existing drugs panobinostat and dexamethasone among patients with relapsed or refractory multiple myeloma. This study will also look at the response and clinical benefit of the treatment and the progression-free survival and overall survival of study participants.

DETAILED DESCRIPTION:
The primary objective of this study is to define the tolerability and safety of MLN9708 (ixazomib) administered on a day 1,8,15 every 28 day schedule up to 4mg in combination with fixed doses of panobinostat and dexamethasone in patients with relapsed or refractory myeloma.

The secondary objectives of this study are to assess response and clinical benefit response rates according to international uniform response criteria and adapted EBMT criteria, respectively. And to assess progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patients must carry a diagnosis of symptomatic multiple myeloma according to international myeloma working group criteria and have relapsed or refractory disease according to international uniform response criteria and must have previously received therapy with a proteasome inhibitor and an IMiD™
* Must have measurable disease defined as any of the following: Serum m-spike ≥ 1g/dL, 24 h urine m-spike of at least 200mg/d, involved serum free light chains ≥ 100mg/L with abnormal serum free light chain ratio, bone marrow plasma cells of at least 30%
* ECOG PS ≤ 2
* No gastro-intestinal condition, that in the opinion of the treating physician or the principal investigator significantly limits oral absorption
* No serious uncontrolled coexisting medical condition
* Patients must meet the following laboratory criteria:

  * ANC ≥ 1.0 x 10^9/L without use of pegfilgrastim in the preceding 21 days and without non-pegylated G-CSF or GM-CSF within 7 days prior to study entry
  * Hemoglobin ≥ 8 g/dl (may be after transfusion of packed red blood cells or use of erythropoiesis stimulating agents)
  * Platelets ≥ 70x 10^9/L without platelet transfusion 7 days prior to study entry
  * AST and ALT ≤ 2.5 x ULN
  * Serum bilirubin ≤ 1.5 x ULN
  * Serum potassium ≥ LLN and serum magnesium ≥ LLN (electrolyte levels may be achieved with repletion or other supportive medications like potassium sparing diuretics)
  * Creatinine clearance ≥ 30 mL/min according to Cockroft-Gault formula
  * Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Baseline MUGA or ECHO must demonstrate LVEF ≥ 45%
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to start of study treatment
* Male patients, even if surgically sterilized (i.e., status post vasectomy), have to either:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study treatment, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.
* Female patients have to fulfill one of the following:

  * Be postmenopausal for at least 1 year before the Screening visit, OR
  * Be surgically sterile, OR
  * If of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study treatment
  * Oral contraceptives are generally metabolized by CYP3A4. Since the induction potential of panobinostat to induce CYP3A4 is unknown, patients who are using oral contraceptives as a method of contraception, and are sexually active, should use another effective contraceptive method, AND Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* At least 7 days must have passed since the last treatment with lenalidomide, pomalidomide, thalidomide, proteasome inhibitors, or low dose cyclophosphamide (up to 50mg daily), at least 21 days must have passed since the last treatment with daratumumab, elotuzumab, investigational therapy and most conventional chemotherapy including cyclophosphamide above 50mg per dose, bendamustine, doxorubicin, cisplatin, and etoposide; and at least 35 days since the last treatment with melphalan.

Exclusion Criteria:

* Prior anti-cancer treatment with MLN9708 (ixazomib), HDAC, DAC, HSP90 inhibitors or valproic acid
* Prior participation in a randomized controlled study that included MLN9708 (ixazomib) in one of the treatment arms independent of whether assigned to MLN9708 (ixazomib) or not
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible)
  * Any history of ventricular fibrillation or torsade de pointes
  * Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
  * Screening ECG with a QTcF > 470 msec (QTcF=QT/3√RR). If potassium or magnesium blood levels are below normal limits, consider repeating ECG after correction of these electrolytes
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
  * Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Impairment of GI function or GI disease that may significantly alter the swallowing absorption of panobinostat and MLN9708
* Patients with diarrhea > CTCAE (version 4.03) grade 2
* Patient has ≥ Grade 3 peripheral neuropathy, or ≥ Grade 2 with pain on clinical examination during the screening period.
* Patients with known metastasis of malignant plasma cells to the central nervous system (if not suspected nonspecific testing is required)
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug. If an alternative medication that does not risk QT prolongation can safely be used in the opinion of the treating physician and the treatment is changed to that medication, the patient may be enrolled.
* Patients who have not passed the nadir of bone marrow suppression from previous anti-myeloma therapy yet. If in doubt, serial CBCs with differential should be obtained.
* The corticosteroids prednisone and dexamethasone may be continued until the day before treatment start if all related adverse events are controlled at CTCAE version 4.03 grade ≤ 1.
* Patients who have received radiation therapy to more than half of the pelvis or more than half of the spine within ≤ 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Systemic treatment, within 14 days before study enrollment, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus hepatitis, or known active hepatitis C virus hepatitis.
* Concurrent diagnosis of another malignancy if either systemic treatment or surgery is expected to be required within 2 years from study entry.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment unless the patient is felt to have fully recovered and any antibiotics that are continued are either beta lactam antibiotics or are specifically allowed on study.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Valent, MD, Principal Investigator — Case Comprehensive Cancer Center; Ehsan Malek, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- DL1 - 3mg Lxazomib; DL2 - 4mg Lxazomib: Panobinostat: 20mg, on day 1, 3, 5, 15, 17, 19, 28 Dexamethasone: 20mg, on day 1, 2, 8, 9, 15, 16, 28 MLN9708: 3mg on day 1, 8, 15, 28
Period: Weeks 1-4
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
Started | 4 (1 extra participant accidentally treated at DL1 (in addition to initial 3).) | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: Phase II Portion of Study at DL2
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
Started | 0 | 9
Completed | 0 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Ixazomib - DL 1
- Phase I/II: Ixazomib -DL2
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase I/II | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 1 | 7 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 11 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 11 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity According to CTCAE Version 4.03
Description: Number of Participants with Dose Limiting Toxicity of MLN9708 (lxazomib) according to CTCAE version 4.03
Time Frame: at 28 days from start of treatment
Population: All participants who received treatment in the phase I portion of the study
Measure: Count of Participants; unit: Participants
Groups:
- Dose Levels 1: Panobinostat: 20mg, on day 1, 3, 5, 15, 17, 19, 28 Dexamethasone: 20mg, on day 1, 2, 8, 9, 15, 16, 28 MLN9708: 3mg on day 1, 8, 15, 28
Arm/Group | Dose Levels 1
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Response to Combination Therapy (Panobinostat, Dexamethasone, MLN9708)
Description: Response to intervention as measured by international uniform response criteria and clinical benefit response according to modified EBMT response criteria, comparing myeloma panels obtained at the beginning of each cycle that include SPEP, 24 h UPEP, serum and urine IFEs, and serum free light chains to results at screening. In addition a baseline bone marrow exam and skeletal survey will be obtained and repeated as clinically indicated and for assessment of complete remission (bone marrow)
Time Frame: 4 months (102 days)
Measure: Number; unit: participants
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
Number analyzed (Participants) | 4 | 12
participants | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be the number of days from study entry to progression or death of any cause, whichever comes first.
  Progression-free survival is survival with absence of progressive disease, defined by
  * An increase of 25% from lowest response value in any one or more of the following:
    * Serum M-component (absolute increase must be >0.5 g/100 ml) *
    * Urine M-component (absolute increase must be >200mg per 24 h)
    * Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be >100 mg/l)
    * Bone marrow plasma cell percentage (absolute % must be >10%)
  * And / or:
    * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
    * Development of hypercalcemia (corrected serum calcium >11.5 mg/100 ml) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: 1 year from start of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
Number analyzed (Participants) | 4 | 12
months | 1.2 [0.7 to 6.0] | 3.5 [0.9 to 7.4]

4. Secondary Outcome: Overall Survival
Description: Overall survival for all will be the number of months from study entry to death from any cause.
Time Frame: up to 3 years from start of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
Number analyzed (Participants) | 4 | 12
months | 12.8 [1.7 to 30.4] | 17.6 [11.9 to 22.9]

ADVERSE EVENTS:
Time Frame: 30 days post last study drug administration
Groups:
- DL2 - 4mg Lxazomib: Panobinostat: 20mg, on day 1, 3, 5, 15, 17, 19, 28 Dexamethasone: 20mg, on day 1, 2, 8, 9, 15, 16, 28 MLN9708: 4mg on day 1, 8, 15, 28
Arm/Group | DL1 - 3mg Lxazomib | DL2 - 4mg Lxazomib
All-Cause Mortality (participants affected / at risk) | 4/4 | 9/12
Serious Adverse Events (participants affected / at risk) | 1/4 | 5/12
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 - 3mg Lxazomib (N=4) | DL2 - 4mg Lxazomib (N=12)
Hyperviscosity (Infections and infestations) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 2
Skin Infection (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 - 3mg Lxazomib (N=4) | DL2 - 4mg Lxazomib (N=12)
anemia (Blood and lymphatic system disorders) | 1 | 4
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 4
Lymphocyte count increased (Blood and lymphatic system disorders) | 0 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 3
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 4
White blood cell decreased (Blood and lymphatic system disorders) | 0 | 3
creatinine increased (Investigations) | 0 | 2
dizziness (Nervous system disorders) | 0 | 2
anorexia (Metabolism and nutrition disorders) | 0 | 2
fever (General disorders) | 0 | 2
edema face (General disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
scalp psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
bruising (Skin and subcutaneous tissue disorders) | 0 | 1
respiratory infection (Infections and infestations) | 1 | 0
headache (Nervous system disorders) | 1 | 2
fatigue (General disorders) | 0 | 3
constipation (Gastrointestinal disorders) | 0 | 2
irritability (General disorders) | 0 | 2
blurred vision (Eye disorders) | 0 | 1
tremors (Nervous system disorders) | 0 | 2
abdominal pain (Gastrointestinal disorders) | 0 | 2
dyspepsia (Gastrointestinal disorders) | 0 | 1
flatulence (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypohosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hemoglobinuria (Renal and urinary disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Breast infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 3 | 6
Taste changes (Gastrointestinal disorders) | 0 | 1
Edema Limbs (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shingles (Infections and infestations) | 0 | 1
Belching (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT02057640/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT02057640/Prot_SAP_001.pdf